CLINICAL TRIAL: NCT01105182
Title: A Prospective Study of Radiofrequency Ablation Combined With Chemotherapy for Pulmonary Tumors
Brief Title: Radiofrequency Ablation Combined With Chemotherapy for Pulmonary Tumors
Acronym: FACPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: The First Affiliated Hospital of Guangzhou Medical College, Guangzhou Medical College
Other Study IDs: FAHG20100201
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2009-12

CONDITIONS: NSCLC; Pulmonary Metastases
Keywords: Radiofrequency Ablation
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Radiofrequency Ablation
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Radiofrequency ablation is an inpatient procedure typically requiring one overnight stay in the hospital.
  Other Names: WHK-3 RFA (Welfare Electronics Co., Beijing PR China)

SUMMARY:
The purpose of this study is to assess short and long term outcomes after radiofrequency ablation (RFA) combined with chemotherapy for pulmonary malignancies in patients who are not candidates for surgical resection. This study will evaluate the efficacy of RFA combined with chemotherapy for the treatment of lung tumors by assessing its impact on local tumor control, progression free survival, overall survival, dyspnea score and quality of life (QOL).

DETAILED DESCRIPTION:
Percutaneous image-guided RFA is a minimally invasive technique used to treat solid tumours. Because of its ability to produce large volumes of coagulation necrosis in a controlled fashion, this technique has gained acceptance as a viable therapeutic option for unresectable liver malignancies. Recently, RFA has been proposed as a viable option for the treatment of pulmonary malignancies. Experimental studies in animal tumor models have confirmed the effectiveness of RFA in the destruction of experimentally-induced pulmonary malignancies. Pilot clinical investigations have suggested that the treatment can achieve high proportions of tumor response. We designed a prospective clinical trial aimed at assessing feasibility, safety and effectiveness of RFA combined with chemotherapy in the treatment of lung malignancies.

ELIGIBILITY:
Inclusion Criteria:

* adult (> 18 years) male or female patient
* patient has biopsy-proven NSCLC or lung metastasis
* patient has been rejected for surgery and has been considered unfit for radiation therapy
* each 6 cm or smaller in greatest diameter of tumor, by CT scan
* tumors are located at least 1 cm from trachea; main bronchi; esophagus; aorta; aortic arch branches; pulmonary artery; and heart
* tumors are accessible by percutaneous route
* patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* patient has platelet count > 100 x 109 /L and international normalized ratio ≤ 1.5
* patient has signed written informed consent prior to any study specific procedures.

Exclusion Criteria:

* patient is considered at high-risk for RF ablation due to major co-morbid medical conditions
* patient has more than 3 tumors / lung
* patient has at least one tumor > 6 cm in greatest diameter
* tumor is associated with atelectasis or obstructive pneumonitis
* patient has renal failure requiring hemodialysis or peritoneal dialysis
* patient has active clinically serious infection
* patient has history of organ allograft
* patient has history of substance abuse or any medical, psychological or social conditions that may interfere with his / her participation in the study or evaluation of the study results
* patient is pregnant or breast-feeding
* patient has ECOG performance status > 2
* patient has platelet count ≤ 100 x 109 /L or international normalized ratio > 1.5.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary malignancies are not candidates for surgical resectionpatients.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 months

SECONDARY OUTCOMES:
Overall survival | 3 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, FACS, Principal Investigator — Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China